CLINICAL TRIAL: NCT03988426
Title: Clinical Phase 3 Study to Evaluate the Efficacy, Tolerability and Safety of Subcutaneous Human Immunoglobulin (Octanorm) in Patients With Primary Immunodeficiency Diseases.
Brief Title: Study to Evaluate the Efficacy, Tolerability and Safety of Octanorm in Patients With Primary Immunodeficiency Diseases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCGAM-04
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-02

CONDITIONS: Primary Immune Deficiency Disorder
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Octanorm (Experimental): Human Normal Immunoglobulin for Subcutaneous Administration (Octanorm) is a liquid formulation of normal human IgG at a concentration of 16.5% administered as a SC infusion at weekly intervals (either done at the study center [during first training sessions and then for every 4th administration] or at home by the patient or caregiver). The initial weekly dose was determined based on subjects' previous IVIG treatment.
  Interventions: Biological: Octanorm

INTERVENTIONS:
Biological: Octanorm — Octanorm

SUMMARY:
Clinical phase 3 study to evaluate the efficacy, tolerability and safety of subcutaneous human immunoglobulin (octanorm) in patients with primary immunodeficiency diseases.

DETAILED DESCRIPTION:
Octanorm (cutaquig®) is a 16.5% human normal immunoglobulin solution developed by Octapharma for subcutaneous administration (SCIG). It is supplied as a liquid formulation ready to use. One important therapeutic use of immunoglobulins is to provide antibodies to prevent viral and bacterial diseases (replacement therapy). Children and adults with a Primary Immunodeficiency Disease (PID) have an increased risk of recurrent bacterial and viral infections. These diseases can be severe and can lead to substantial morbidity. Responses to antibacterial therapy are often poor. At present, most primary immune deficiencies are not curable, but SCIGs have been shown to decrease the total number of severe infections and the duration of hospitalization. This study evaluated the efficacy, safety and tolerability of octanorm in adult PID patients in an open-label, multi center, phase 3 study with an 8-week wash-in/wash-out period followed by a 6-month efficacy period

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥18 years and ≤70 years.
2. Confirmed diagnosis of PI requiring immunoglobulin replacement therapy due to hypogammaglobulinaemia or agammaglobulinaemia. The type of PI should be recorded.
3. Patients with at least 4 infusions on regular treatment with any Intravenous Immunoglobulin (IVIG) prior to entering the study. Constant IVIG dose between 200 and 800 mg/kg body weight (the individual doses of the last 4 infusions should not vary by more than ±25% of the mean dose for the last 4 infusions).
4. Availability of at least 2 IgG trough levels with an IgG level of ≥5.0 g/L from the period of the last 4 IVIG infusions.
5. Negative result on a pregnancy test (Human Chorionic Gonadotrophin [HCG]-based assay in urine) for women of childbearing potential and use of a reliable method of contraception for the duration of the study. Women of non-childbearing potential must be post-menopausal (amenorrhoeic for at least 12 months) or surgically sterile.

   Examples for medically acceptable methods of birth control for this study include:
   * Oral, implantable, transdermal or injectable contraceptives
   * Intrauterine device
   * Condoms; diaphragm or vaginal ring with spermicidal jellies or cream
   * Sexual abstinence
   * Vasectomised partner
6. Patient must freely give written informed consent.
7. Willingness to comply with all aspects of the protocol, including blood sampling, for the duration of the study.

Exclusion Criteria:

1. Acute infection requiring intravenous (IV) antibiotic treatment within 2 weeks prior to and during the screening period.
2. Known history of adverse reactions to Immunoglobulin A in other products.
3. Patients with body mass index >40 kg/m2
4. Exposure to blood or any blood product or plasma derivatives, other than IVIG treatment of PI, within the past 3 months prior to first infusion of octanorm.
5. Ongoing history of hypersensitivity or persistent reactions to blood or plasma derived products, or any component of the investigational medicinal product (IMP) (such as Polysorbate 80).
6. History of malignancies of lymphoid cells and immunodeficiency with lymphoma.
7. Severe liver function impairment (ALAT 3 times above upper limit of normal).
8. Known protein-losing enteropathies or proteinuria.
9. Presence of renal function impairment (creatinine >120 µM/L or creatinine >1.35 mg/dL), or predisposition for acute renal failure (e.g., any degree of pre-existing renal insufficiency or routine treatment with known nephritic drugs).
10. Treatment with enteral or parenteral steroids for ≥30 days or when given intermittently or as bolus, at daily doses ≥0.15 mg/kg. Inhaled corticosteroids are allowed.
11. Patients with chronic obstructive pulmonary disease (COPD) stage Global Initiative for Chronic Obstructive Lung Disease (GOLD) III or IV.
12. Treatment with immunosuppressive drugs.
13. Live viral vaccination (such as measles, rubella, mumps and varicella) within the last 2 months prior to first infusion of octanorm.
14. Treatment with any IMP within 3 months prior to first infusion of octanorm.
15. Presence of any condition that is likely to interfere with the evaluation of study medication or satisfactory conduct of the trial.
16. Known or suspected to abuse alcohol, drugs, psychotropic agents or other chemicals within the past 12 months prior to first infusion of octanorm.
17. Known or suspected human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infection.
18. Pregnant or nursing women; planned pregnancy during course of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2018-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Toeglhofer, MD, Study Director — Octapharma
Locations (5):
- Russia (5):
  - The State Research Center, Institute of Immunology of the Federal Medical-Biological Agency, Moscow
  - Federal Research Center of Pediatric Hematology, Oncology and Immunology of the Ministry of Health and Social Development of the Russian Federation, Moscow
  - State Medical University, Rostov
  - Pasteur Institute, Saint Petersburg
  - Institute of Immunology and Physiology of the Ural Branch of the Russian Academy of sciences, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Latysheva E, Rodina Y, Sizyakina L, Totolian A, Tuzankina I. Efficacy and safety of octanorm (cutaquig(R)) in adults with primary immunodeficiencies with predominant antibody deficiency: a prospective, open-label study. Immunotherapy. 2020 Apr;12(5):299-309. doi: 10.2217/imt-2020-0012. Epub 2020 Mar 26. PMID 32212944

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants Administered Octanorm: All patients in the study received Octanorm as study drug. Dosage of octanorm was based on the previous dosage of IVIG for each patient: by dividing the previous IVIG dosage by the number of weeks between IVIG administrations. Octanorm was to be administered every week (+/- 2 days) as subcutaneous administration. Administration were either done at the study site (for the first training sessions and then every 4th infusions) or at home (administered by the patient or a caregiver)
Period: Overall Study
Arm/Group | Participants Administered Octanorm
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Full analysis set (FAS population) included all patients who received at least one administration of the study drug and for whom any post-baseline data was available
Arm/Group | All Patients
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 35.24 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Russia | 25
Height [Mean (Standard Deviation); unit: centimeters] | 170 (8.68)
Weight [Mean (Standard Deviation); unit: kilograms] | 66.49 (10.54)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] | 23.02 (3.48)

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Bacterial Infections Per Person-Year on Treatment
Description: Serious Bacterial Infections defined as bacteraemia/sepsis, bacterial meningitis, osteomyelitis/septic arthritis, bacterial pneumonia, and visceral abscess
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Number; unit: SBI per patient year
Arm/Group | Octanorm
Number analyzed (Participants) | 24
SBI per patient year | 0

2. Secondary Outcome: Number of Patients With Other Infections
Description: The number of patients with all infections of any kind or seriousness.
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Octanorm
Number analyzed (Participants) | 24
Participants
  Number of Patients With Infections | 14
  Number of Patients with 0 Infections | 10
  Number of Patients with 1 Infection | 9
  Number of Patients with 2 Infections | 2
  Number of Patients with 3 Infections | 0
  Number of Patients with 4 Infections | 2
  Number of Patients with 5 Infections | 1

3. Secondary Outcome: Number of Other Infections
Description: For other infections, the Medical Dictionary for Regulatory Activities (MedDRA) preferred term was used to determine the type of infection. They were grouped into the following categories as determined by a medical expert: Ear infections, eye infections, infections of the gastrointestinal tract, infections of the genitourinary tract, upper respiratory tract infections, lower respiratory tract infections, infections of the skin, and infections not elsewhere classified.
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Number; unit: Infections
Groups:
- All Patients: Full analysis set
Arm/Group | All Patients
Number analyzed (Participants) | 24
Infections
  Number of Mild Infections | 17
  Number of Moderate Infections | 9
  Number of Severe Infections | 0

4. Secondary Outcome: Time to Resolution of Infections
Description: Since infections were reported as adverse events, the time to resolution of an infection was the time from the start date of the infection adverse event to the end date of the infection adverse event.
Time Frame: Primary Treatment Period (24 Weeks) and Whole Treatment Period (up to 36 Weeks)
Measure: Number; unit: days
Arm/Group | Octanorm
Number analyzed (Participants) | 24
days
  Primary Treatment Period | 9.53
  Whole Treatment Period | 10.32

5. Secondary Outcome: Number of Participants Using Antibiotics From 0 to > 20 Days
Description: Number of patients using antibiotics during the whole treatment period (36 weeks) grouped per number of days with antibiotic usage.
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Octanorm
Number analyzed (Participants) | 24
Participants
  Patients with 0 Treatment Days | 14
  Patients with 5 Treatment Days | 2
  Patients with 7 Treatment Days | 1
  Patients with 8 Treatment Days | 2
  Patients with >20 Treatment Days | 5

6. Secondary Outcome: Annual Rate of Antibiotic Use
Description: The number of antibiotic treatment episodes per person-year of treatment was calculated by the following formula: Total number of antibiotic treatment episodes / patient-years of Octanorm treatment
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Number; unit: treatment episodes per person-year
Arm/Group | Octanorm
Number analyzed (Participants) | 24
treatment episodes per person-year | 1.73

7. Secondary Outcome: Hospitalizations Due to Infection
Description: Number of days spent in hospital due to infection
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Octanorm
Number analyzed (Participants) | 24
days | 0 (0)

8. Secondary Outcome: Rate of Hospitalizations Due to Infection
Description: Annual Rate of Hospitalizations due to Infection
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Number; unit: hospitalizations/person-year
Arm/Group | Octanorm
Number analyzed (Participants) | 24
hospitalizations/person-year | 0

9. Secondary Outcome: Episodes of Fever
Description: Number of episodes of fever
Time Frame: Primary Treatment Period (24 Weeks) and Whole Treatment Period (up to 36 Weeks)
Measure: Number; unit: episodes of fever
Arm/Group | Octanorm
Number analyzed (Participants) | 24
episodes of fever
  Primary Treatment Period | 6
  Whole Treatment Period | 8

10. Secondary Outcome: Rate of Episodes of Fever
Description: The number of episodes of fever per person-year of treatment was calculated by the following formula: Total number of episodes of fever / patient-years of Octanorm treatment
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Number; unit: episodes of fever per person-year
Arm/Group | Octanorm
Number analyzed (Participants) | 24
episodes of fever per person-year | 0.55

11. Secondary Outcome: Patients With Days Missed From Work/Study Due to Infections and Treatment
Description: Total number of patients who missed days from work or study due to infections or treatment thereof.
Time Frame: Primary Treatment Period (24 Weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Octanorm
Number analyzed (Participants) | 24
Participants | 3

12. Secondary Outcome: Changes in the Subscales of the Form-36 Health Survey Scores From Baseline to the End of the Study
Description: The SF-36-HS consists of 36 items organized into 8 subscales. The 8 subscales could be combined into 2 summary scores, physical and mental. The calculated summary scores were transformed to a range of 0-100, where a higher score indicates better health. A positive change score indicates improvement.
Time Frame: Baseline to the end of study (up to 36 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Full Analysis Set: All participants who received at least 1 complete treatment with Octanorm and for whom any post-baseline data was available.
Arm/Group | Full Analysis Set
Number analyzed (Participants) | 25
score on a scale
  Physical Functioning | 2.5 (12.25)
  Role Physical | 8.07 (25.83)
  Bodily Pain | 21.38 (28.12)
  General Health | -1.08 (15.16)
  Vitality | 5.73 (17.67)
  Social Functioning | 7.81 (23.26)
  Role Emotional | 10.76 (22.18)
  Mental Health | 5.83 (20.62)

13. Secondary Outcome: Trough Levels of Serum Total IgG
Description: Total IgG trough concentrations were measured in serum samples taken before each infusion given at the study site.
Time Frame: At baseline and at last infusion (week 33)
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Octanorm
Number analyzed (Participants) | 25
g/L
  Screening Draw 1 | 8.71 (2.68)
  Week 33 | 9.99 (1.79)

14. Secondary Outcome: Number of Participants Experiencing Treatment-Emergent AEs
Description: TEAEs were classified as temporally associated if the onset was during the infusion or within 72 hours after the end of the infusion.
Time Frame: Up to 36 weeks
Measure: Number; unit: patients
Arm/Group | Octanorm
Number analyzed (Participants) | 25
patients
  Without Infusion Site Reactions and With Infection | 18
  Without Infusion Site Reactions/Without Infection | 11
  Infections (only) | 16

15. Secondary Outcome: Proportion of Infusions With at Least 1 Temporally Associated AE
Description: The proportion of infusions with at least 1 temporally associated AE (TAAE) was calculated by dividing the total number of TAAE by the total number of infusions.
Time Frame: Up to 36 weeks
Measure: Number; unit: proportion of infusions
Arm/Group | Octanorm
Number analyzed (Participants) | 25
proportion of infusions | .013

16. Secondary Outcome: Total Number of Adverse Events Regardless of Causality
Description: An AE is any untoward medical occurrence in a study patient receiving an IMP and which does not necessarily have a causal relationship with this treatment.
Time Frame: Up to 36 weeks
Measure: Number; unit: adverse events
Arm/Group | Octanorm
Number analyzed (Participants) | 25
adverse events | 59

17. Secondary Outcome: Number of Related Adverse Events
Description: A related adverse event is an AE for which a causal relationship between the IMP and the AE cannot be ruled out.
Time Frame: Up to 36 weeks
Measure: Number; unit: related adverse events
Arm/Group | Octanorm
Number analyzed (Participants) | 25
related adverse events | 3

18. Secondary Outcome: Number of Infusions With Infusion Site Reaction
Description: Total number of infusions that triggered an infusion site reaction and number of infusions that triggered mild, moderate, severe or no infusion site reactions.
Time Frame: Up to 36 weeks
Measure: Number; unit: infusions
Arm/Group | Octanorm
Number analyzed (Participants) | 25
infusions
  Infusions with Mild Local Site Reactions | 102
  Infusions with Moderate Local Site Reactions | 17
  Infusions with Severe Local Site Reactions | 0
  Infusions with No Infusion Site Reaction | 659

19. Secondary Outcome: Annual Rate of Infections
Description: The annual rate of all infections of any kind of seriousness
Time Frame: Up to 36 weeks
Measure: Number; unit: infections/person-year
Arm/Group | All Patients
Number analyzed (Participants) | 24
infections/person-year | 2.37

ADVERSE EVENTS:
Time Frame: Up to 36 weeks
Arm/Group | Octanorm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 18/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octanorm (N=25)
Dizziness (Nervous system disorders) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 2 (2)
Condition Aggravated (General disorders) | 5 (6)
Respiratory Tract Infection (Infections and infestations) | 6 (8)
Bronchitis (Infections and infestations) | 4 (5)
Rhinitis (Infections and infestations) | 2 (2)
Pharyngitis (Infections and infestations) | 2 (2)
Blood and Lymphatic Infection (Blood and lymphatic system disorders) | 2 (2)
Investigations (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-11-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT03988426/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT03988426/SAP_001.pdf